CLINICAL TRIAL: NCT03823547
Title: Future Optimal Research and Care Evaluation: On the Way to "Personalized Medicine" With an Ongoing Registry of Patients in Daily Clinical Practice (Hart Beter/ FORCE-ACS)
Brief Title: Future Optimal Research and Care Evaluation
Acronym: FORCE-ACS
Status: Recruiting | Type: Observational
Sponsor: J.M. ten Berg (Other)
Collaborators: Vereniging Hart-Beter (Unknown); St. Antonius Hospital (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, J.M. ten Berg, Principle investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Other Study IDs: Hart Beter/FORCE-ACS
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: DAPT; Dual Antiplatelet Therapy; Myocardial infarction; Acute Coronary Syndrome; Ticagrelor; Prasugrel; Clopidogrel; Thrombosis; Myocardial Ischemia; Platelet aggregation inhibitors; Risk scores; Cardiovascular diseases
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Thrombosis; Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Acute coronary syndrome (ACS) is the leading cause of death worldwide. To improve cardiovascular care, research is needed. Current guidelines are mainly based on well controlled RCT's, though evaluation of the impact of such RCT's in the real world is missing. In order to evaluate the impact and to overcome certain limitations of RCT's, a more practical approach is required. In this sense the use of nonrandomized observational studies is an important tool for determining the effectiveness of a therapy in routine clinical practice. One way to gain insight in characteristics of patients presenting in daily clinical practice, is to simply register these characteristics in a prospective manner with adequate follow up.

Objective: To create an ongoing registry for evaluation of clinical long-term impact of diagnostics, various treatments and devices used for ACS, for research and evaluation of quality of care and to evaluate and improve regional quality of care and cooperation between PCI and non-PCI centers.

DETAILED DESCRIPTION:
Rationale:

Acute coronary syndrome (ACS) is the leading cause of death worldwide. To improve cardiovascular care, research is needed. Current guidelines are mainly based on well controlled RCT's, though evaluation of the impact of such RCT's in the real world is missing. Different clinical settings, non-ideal therapy adherence and broader patient populations in the real world than those studied in traditional RCTs may however provide different results. Furthermore, RCTs are intrinsically limited to answer questions about a specific population of interest, require substantial resource investments and may have limitations in investigating certain issues for ethical reasons.

In order to evaluate the impact and to overcome certain limitations of RCT's, a more practical approach is required. In this sense the use of nonrandomized observational studies is an important tool for determining the effectiveness of a therapy in routine clinical practice. One way to gain insight in characteristics of patients presenting in daily clinical practice, is to simply register these characteristics in a prospective manner with adequate follow up. These characteristics may include clinical parameters but also possibly genetic information. Such a detailed registry is now possible due to improvements in information technology, as electronic patient records permit more (semi-) automatic and uniform capture of clinical parameters and outcomes. While observational studies may often be limited in their ability to account for confounding and bias due to patient selection, recent evidence has shown that by careful use of advanced statistical analytical methods and open reporting paradigms the quality of the level of evidence is excellent.

Objectives:

1. To create a database for future research, especially in the view of personalized medicine, and quality of care.
2. To evaluate clinical long-term impact of medication, devices and diagnostic tools used for patients with an ACS.
3. To test the efficacy and safety of any new drug/device versus the current treatment and the results of any drug/device in daily practice versus in trials
4. To evaluate routine follow-up and current health-care pathways in patients with acute coronary syndrome in the Dutch healthcare system in terms of mortality, recurrent ischemic events, recurrent hospital admissions and quality of life
5. To evaluate the use of risk scores (e.g. PRECISE-DAPT score, DAPT-score) to define the optimal duration of antiplatelet drugs
6. To evaluate follow-up of patients referred to general practitioners as compared to of patients continued to be treated by cardiologists
7. To increase adherence to current guidelines, taking into account the ongoing improvements of modern patient care and future changes of treatment guidelines in patients with ACS in order to improve secondary prevention in terms of reducing recurrent ischemic events and preventing adverse outcomes, such as bleeding

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with ACS
* Age ≥ 18 years

Exclusion Criteria:

* No oral or signed informed consent available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the hospital ward with acute coronary syndrome or symptoms suggestive for acute coronary syndrome are invited to participate in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2050-06-30 (Estimated); Study Completion 2050-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with | 3 years
  * All-cause mortality
  * Myocardial infarction
  * Stent thrombosis
  * Stroke
  * Revascularisation
  * All bleeding requiring medical evaluation

SECONDARY OUTCOMES:
Number of participants with | 3 years
  * mortality classification into cause-of-death (i.e cardiovascular, cardiac, vascular, cerebrovascular, death due to bleeding)
  * bleeding classification according to different bleeding criteria (i.e. TIMI, BARC, GUSTO, PLATO)
  * cessation (and duration) of antiplatelet therapy after ACS
  * patient related outcome measures, as reported in quality of life questionnaires (e.g. SF-12, Seattle Angina Questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Dekker, Drs., Study Chair — St. Antonius Hospital
Locations (4):
- Netherlands (4):
  - Gelre Ziekenhuizem, Apeldoorn, Gelderland
  - Rijnstate Arnhem, Arnhem, Gelderland
  - Gelderse Vallei, Ede, Gelderland
  - Ziekenhuis Rivierenland, Tiel, Gelderland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van den Broek WWA, Azzahhafi J, Chan Pin Yin DRPP, van der Sangen NMR, Sivanesan S, Dijksman LM, Walhout RJ, Tjon Joe Gin M, Breet NJ, Langerveld J, Vlachojannis GJ, van Bommel RJ, Appelman Y, van Schaik RHN, Henriques JPS, Kikkert WJ, Ten Berg JM. Cost-effectiveness of implementing a genotype-guided de-escalation strategy in patients with acute coronary syndrome. Eur Heart J Cardiovasc Pharmacother. 2025 May 2;11(3):230-240. doi: 10.1093/ehjcvp/pvae087. PMID 39537191
- [Derived] van der Sangen NMR, Azzahhafi J, Chan Pin Yin DRPP, Peper J, Rayhi S, Walhout RJ, Tjon Joe Gin M, Nicastia DM, Langerveld J, Vlachojannis GJ, van Bommel RJ, Appelman Y, Henriques JPS, Ten Berg JM, Kikkert WJ. External validation of the GRACE risk score and the risk-treatment paradox in patients with acute coronary syndrome. Open Heart. 2022 Mar;9(1):e001984. doi: 10.1136/openhrt-2022-001984. PMID 35354660
- [Derived] Chan Pin Yin DRPP, Vos GA, van der Sangen NMR, Walhout R, Tjon Joe Gin RM, Nicastia DM, Langerveld J, Claassens DMF, Gimbel ME, Azzahhafi J, Bor WL, Oirbans T, Dekker J, Vlachojannis GJ, van Bommel RJ, Appelman Y, Henriques JPS, Kikkert WJ, Ten Berg JM. Rationale and Design of the Future Optimal Research and Care Evaluation in Patients with Acute Coronary Syndrome (FORCE-ACS) Registry: Towards "Personalized Medicine" in Daily Clinical Practice. J Clin Med. 2020 Sep 30;9(10):3173. doi: 10.3390/jcm9103173. PMID 33007932